CLINICAL TRIAL: NCT00161798
Title: Double-blind, Randomized, Multicenter Dose-finding Study to Investigate the Safety and Immunogenicity of Two Vaccinations With FSME IMMUN NEW in Healthy Volunteers Aged 6 to 16 Years.
Brief Title: Dose-finding Study to Investigate the Safety and Immunogenicity of Two Vaccinations With FSME IMMUN NEW in Healthy Volunteers Aged 6 to 16 Years.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 205
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Tick-borne Encephalitis
MeSH Terms: conditions — Encephalitis, Tick-Borne

INTERVENTIONS:
Biological: Tick-borne encephalitis vaccine

SUMMARY:
The purpose of this study is to investigate the safety and immunogenicity of three different concentrations of a TBE vaccine will be investigated in healthy children aged 6 to 16 years.

ELIGIBILITY:
Inclusion Criteria:

Male and female children will be eligible for participation in this study if:

* they are 6 years (from the 6th birthday) to 16 years old (to the last day before the 16th birthday);
* they are clinically healthy;
* their legal representative - and if older than 8 years the volunteer - understands the nature of the study, agrees to its provisions and gives written informed consent;
* their legal representative agrees to keep a Volunteer Diary.

For safety reasons female volunteers capable of bearing children have to fulfill the following inclusion criteria at study start:

* negative pregnancy test at study start;
* they agree to employ adequate birth control measures for the duration of the study.

Exclusion Criteria:

Children will be excluded from participation in this study if they:

* have a history of any previous TBE vaccination;
* have a history of TBE infection or show evidence of a latent TBE infection (as demonstrated by screening ELISA > 126 VIEU/ml and / or neutralization test > 1:10);
* have a history of allergic reactions, in particular to one of the components of the vaccine;
* have received antipyretics within 4 hours prior to the first TBE vaccination;
* suffer from a disease that cannot be effectively treated or stabilized;
* suffer from a disease (e.g. autoimmune disease) or are undergoing a form of treatment that can be expected to influence immunological functions;
* suffer from chronic, degenerative and / or inflammatory disease of the central nervous system;
* are known to be HIV positive (a special HIV test is not required for the purpose of the study);
* suffer from a febrile illness at study entry;
* have a history of vaccination against yellow fever and / or Japanese B-encephalitis;
* are participating simultaneously in another clinical trial.
* if female, are pregnant or breast feeding

Volunteers who meet the inclusion / exclusion criteria, but have a febrile illness (body temperature >= 38° C, measured orally) at the scheduled time of vaccination, will not be vaccinated before their body temperature returns to normal.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Dates: Start 2001-09; Study Completion 2002-03

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Behre, MD, Principal Investigator — Hauptstrasse 240, 77694 Kehl, Germany
Locations (23):
- Germany (23):
  - Neuschwansteinstrasse 5, Augsburg
  - Marktplatz 33, Bad Saulgau
  - Hauptstrasse 9, Bietigheim-Bissingen
  - Salzgasse 11, Calw
  - Mohrenstrasse 8, Coburg
  - Bahnhofstrasse 1, Elzach
  - Rheinstrasse 13, Ettenheim
  - Peter-Seifert Strasse 5, Gersfeld
  - Solothurner Strasse 2, Heilbronn
  - Hauptstraße 240, Kehl
  - Schwarzwaldstrasse 20, Kirchzarten
  - Altoettingerstrasse 3, Landsberg
  - Rastatter Strasse 7, Mannheim-Secken
  - Wilhelmstrasse 25, Metzingen
  - Heubischer Strasse 39, Neustadt/Cbg
  - Dohmbuehlerstrasse 8, Nuremberg
  - Schwarzwaldstrasse 18, Oberkirch
  - Wilhelmstrasse 7, Offenburg
  - Asternweg 11a, Offenburg
  - Bergstrasse 27, Rottweil
  - Berneckstrasse 19, Schrammberg
  - Hauptstrasse 11, Tegernsee
  - Broner Platz 6, Weingarten